CLINICAL TRIAL: NCT06274684
Title: Feasibility of Virtual Reality Assistance in Prostate Biopsy Under Local Anesthesia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Sylvain Vanoli, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01100
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Virtual Reality; VR; Anxiety; Prostate biopsies; Transperineal biopsies
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality assistance group (Experimental): Patient receiving VR headset during prostate biopsies
  Interventions: Device: Use of Virtual Reality Assistance during prostate biopsies
- Control group (No Intervention)

INTERVENTIONS:
Device: Use of Virtual Reality Assistance during prostate biopsies — Patient will be equipped with VR headset providing a immersive experience during prostate biopsies
  Arms: Virtual Reality assistance group

SUMMARY:
The goal of this clinical trial is to test the impact of Virtual Reality (VR) assistance for anxiety management of patients undergoing prostate biopsies in local anaesthesia.

The main question it aims to answer:

- Is there a significant decrease on anxiety level thanks to VR-assistance?

Participants will be equipped with VR headset providing an immersive visual experience accompanied with a hypnoses oriented audio during the entire procedure.

Researchers will compare standardised anxiety scores with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Indication for prostate biopsies
* Informed consent

Exclusion Criteria:

* Local anaesthesia contra-indication (allergy)
* Claustrophobia
* Major cognitive impairment and impossibility of answering the standardised questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-19 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | On the day of the biopsies (before the procedure) and one day after procedure
  State-Trait Anxiety Inventory (STAI) validated questionnaires

SECONDARY OUTCOMES:
Anxiety level of the surgeon | One day after procedure
  Short-Form State-Trait Anxiety Inventory validated questionnaires
Biopsies complications | In the 30 days following prostate biopsies